CLINICAL TRIAL: NCT00378729
Title: PERCING : Ovarian Drilling Versus Ovarian Stimulation + Intra Uterine Insemination (IUI) + Metformin in the PCOS (PolyCystic Ovaries Syndrome) Treatment
Brief Title: Surgical Ovarian Drilling Versus Hormonal Treatment for Infertility Associated to PolyCystic Ovaries Syndrome (PCOS)
Acronym: PERCING
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hopital Antoine Beclere (Other); Hôpital Jean Verdier (Other); Jean Rostand Intercommoned Hospital (Unknown); Centre Hospitalier Universitaire, Amiens (Other); University Hospital, Caen (Other); University Hospital, Clermont-Ferrand (Other); Lille Hospital : Jeanne de Flandre Hospital (Unknown); University Hospital, Strasbourg, France (Other); CMCO SIHCUS, Schiltingheim (Other); Study and research center of sterility (Lyon) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051008
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; FERTILOSCOPY; Ovarian hyperstimulation; Multiple pregnancies; Patient with PCOS (Rotterdam criteria); Failure of treatment with Clomiphene Citrate; Age between 18 and 36 years old; Spermogram must be normal; Permeability of Fallopian tubes
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Metformin and FSHr
- B (Active Comparator)
  Interventions: Procedure: Ovarian drilling by FERTILOSCOPY

INTERVENTIONS:
Drug: Metformin and FSHr — treatment for infertility
  Other Names: treatment for infertility
  Arms: A
Procedure: Ovarian drilling by FERTILOSCOPY — surgical ovarian drilling
  Other Names: surgical ovarian drilling
  Arms: B

SUMMARY:
PolysCsytic Ovaries Syndrome (PCOS) is the most frequent endocrinopathy. The first stage of infertility treatment is Clomiphene Citrate which leads to 50 % pregnancies. In case of failure, it is possible to propose surgical ovarian drilling or ovarian hyperstimulation with Intra Uterine Insemination (IUI) which lead to 50% pregnancies each. However, surgical treatment could be associated to surgical complications, and medical treatment could be associated to ovarian hyperstimulation syndrome and/or multiple pregnancies.

The aim of this study is to compare the two treatments to demonstrate the equivalence of efficacy and the diminution of multiple pregnancies by the surgical treatments. After an ambulatory surgery we will observe the spontaneous fertility during 9 months. For the medical treatment, Metformin is proposed during 9 months associated with 3 cycles of ovarian hyperstimulation and IUI if the sperm is normal

DETAILED DESCRIPTION:
PolysCsytic Ovaries Syndrome (PCOS) is the most frequent endocrinopathy. The first stage of infertility treatment is Clomiphene Citrate which leads to 50 % pregnancies. In case of failure, it is possible to propose surgical ovarian drilling or ovarian hyperstimulation with Intra Uterine Insemination (IUI) which lead to 50% pregnancies each. However, surgical treatment could be associated to surgical complications, and medical treatment could be associated to ovarian hyperstimulation syndrome and/or multiple pregnancies.

The aim of this study is to compare the two treatments to demonstrate the equivalence of efficacy and the diminution of multiple pregnancies by the surgical treatments. After an ambulatory surgery we will observe the spontaneous fertility during 9 months. For the medical treatment, Metformin is proposed during 9 months associated with 3 cycles of ovarian hyperstimulation and IUI if the sperm is normal Ovarian drilling will be performed by FERTILOSCOPY. 126 patients will be necessary in each group (with interval of equivalence : 10%).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 36 years old
* Female patient with PCOS (Rotterdam criteria)
* Failure of treatment with Clomiphene Citrate
* Informed consent
* Female patient with medical assurance
* Patient in failure with PCOS and Clomiphene citrate

Exclusion Criteria:

* Female patient is over 36 years old
* Thyroid disease (4<TSH<0.3 mUI/L)
* Virilizing tumor
* FERTILOSCOPY non possible (Douglas cul de sac clinically fixed)
* Anormality of SPERMOGRAM (abnormal time of migration of survival)
* Prolactin > 1.5 N
* Anormality of 17-OH Progesterone (<2 ng/mL)
* Fallopian tubes non permeable TMS< 5 Millions
* Female patient participant or have been participated to another clinical trial during the last month before the inclusion
* Female patient without medical assurance

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the cumulative rate of on-going pregnancy (>12 weeks of amenorrhoea) obtained during 9 months of follow-up | during 9 months of follow-up

SECONDARY OUTCOMES:
Evaluation of tolerance | during the study
Occurrence of multiple pregnancies | at the end of the study
Duration of the menstrual cycles and hormonal ovarian dosages | during the study
Occurrence of spontaneous miscarriages | at the end of the study
Body Mass Index with each visit | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Hervé FERNANDEZ, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Antoine Beclere, Clamart, France

REFERENCES:
- [Background] Fernandez H, Watrelot A, Alby JD, Kadoch J, Gervaise A, deTayrac R, Frydman R. Fertility after ovarian drilling by transvaginal fertiloscopy for treatment of polycystic ovary syndrome. J Am Assoc Gynecol Laparosc. 2004 Aug;11(3):374-8. doi: 10.1016/s1074-3804(05)60054-0. PMID 15559352